CLINICAL TRIAL: NCT05132699
Title: Enhancing Prolonged Exposure With Cannabidiol to Treat Posttraumatic Stress Disorder: A Pilot Study
Brief Title: Enhancing Prolonged Exposure With Cannabidiol to Treat Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Casey Straud, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20210711H; UL1TR002645 (NIH); KL2TR002646 (NIH)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Posttraumatic Stress Disorder; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cannabidiol; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled clinical trial. Permuted block randomization will ensure equal allocation of participants to either study drug or placebo. Randomization will be performed by a designated study team member.
Who Masked: Participant, Investigator
Masking Description: A compounding pharmacy will supply both the study drug and a matching strawberry flavored liquid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cannabidiol (CBD) (Active Comparator): Epidiolex oral solution 500mg (5ml) per day
  Interventions: Drug: Cannabidiol (CBD) oral solution; Behavioral: Massed Prolonged Exposure (mPE)
- Placebo (Placebo Comparator): Placebo oral solution 5ml per day
  Interventions: Drug: Placebo; Behavioral: Massed Prolonged Exposure (mPE)

INTERVENTIONS:
Drug: Cannabidiol (CBD) oral solution — An oral strawberry flavored liquid, taken as a 2.5ml (250mg) dose twice a day
  Other Names: Epidiolex
  Arms: Cannabidiol (CBD)
Drug: Placebo — An inert strawberry flavored oral solution, taken as a 2.5ml dose twice a day
  Other Names: Placebo oral solution
  Arms: Placebo
Behavioral: Massed Prolonged Exposure (mPE) — mPE, delivered daily Monday through Friday over two weeks, utilizes exposure-based interventions to target psychological mechanisms (i.e., experiential and behavioral avoidance; maladaptive cognitive changes) that are thought to maintain trauma-related symptoms.
  Other Names: Behavioral Therapy

SUMMARY:
The primary goal of this pilot project is to demonstrate the safety and feasibility of using Cannabidiol (CBD) in combination with standard of care prolonged exposure (PE) psychotherapy to reduce PTSD symptoms.

DETAILED DESCRIPTION:
This study is an early Phase II double-blind, pilot randomized controlled clinical trial. The study team will use a permuted block randomization design stratified by a Posttraumatic Stress Disorder (PTSD) severity median score on the PTSD Checklist (PCL-5) derived from a recently completed STRONG STAR repository. Participants will be up to 24 individuals with PTSD to investigate the safety, feasibility, and PTSD symptom change associated with CBD 250mg taken twice a day for 18 days (n=up to 12) vs. placebo (n=up to12) in combination with a standard of care, 10-sessions massed PE psychotherapy administered over 2 weeks. Aims 2 and 3 will evaluate biochemical and physiological outcomes associated with the brain endocannabinoid (eCB) and PTSD that may be affected by CBD. Permuted block randomization is advantageous in small clinical trials to ensure equal allocation of participants in each condition. Participant randomization will be subdivided into randomized blocks of four, two patients in each block will be assigned to CBD and two will be assigned to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the age of 18 to 65 years old at time of screening.
2. Able to write, read, and speak English
3. PTSD diagnosis as assessed by Clinician-Administered Posttraumatic Stress Scale (CAPS-5)
4. Stable medication regimen for at least four weeks prior to the onset of study participation.

Exclusion Criteria:

1. History of opiate, cocaine, methamphetamine, benzodiazepine, or cannabis abuse as determined by the National Institute of Drug Abuse Quick Screen (NIDA-Q).
2. Currently using opiates, cocaine, methamphetamines, benzodiazepines, or cannabis as evidenced by a positive urine drug screen prior to enrollment.
3. Currently pregnant as determined by a positive urine pregnancy test prior to enrollment.
4. Current clinically significant alcohol abuse in the past two weeks on the Quick Drinking Screen (QDS).
5. Currently breastfeeding.
6. Ongoing illness or physical health problem(s) that may be exacerbated by CBD (e.g., history of liver problems)
7. History of significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to cannabinoids.
8. Concomitant medications with possible CBD-drug interactions
9. Alanine transaminase (ALT) or Aspartate transaminase (AST) enzyme levels 3x normal limits.
10. Concurrent engagement in trauma-related psychotherapy for PTSD.
11. Current or past DSM-5 diagnosis of psychotic disorder or bipolar disorder as determined on the Mini International Neuropsychiatric Interview (MINI 7.0).
12. Suicide attempt in the last year and/or suicide risk requiring immediate intervention or requiring a higher level of care than can be provided by the study treatment as determined by the Self-Injurious Thoughts and Behaviors Interview (SIT-BI).
13. Allergy to sesame seed oil.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey Straud, PsyD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio - STRONG STAR Northwest Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A STRONG STAR Institutional Review board (IRB) approved Repository to enable the STRONG STAR Consortium to store specimens and data for future use. Study databases are established and maintained by the STRONG STAR Data and Statistics Services. All Repository data will be identified with a different code number that can be cross linked to the original study code only through records maintained by the STRONG STAR Data and Statistics Services. At the conclusion of this study, participants who signed the consent to have their data placed in the STRONG STAR Repository will be maintained under the UT Health San Antonio IRB-approved Repository protocol. For participants who decline participation in the STRONG STAR Repository, their data will be de-identified, and the data maintained in the Repository without identifiers.
  Summary results will also be shared on ClincalTrials.gov.
Supporting Information: Study Protocol, SAP
Time Frame: After study enrollment is closed and data analysis is complete. Data will be stored in the repository and accessible as long as the IRB approval for this data base remains current.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol (CBD) | Placebo
Started | 11 | 10
Completed | 8 | 10
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: 21 were randomized into CBD (n=11) or placebo (n=10).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol (CBD) | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 21 were randomized into CBD (n=11) or placebo (n=10). 1 individual in the placebo condition was not included in analyses (A PI drop due to participant non-compliance and loss of eligibility. Data gathered from this participant was not evaluable).
  years | 45.9 (12.2) | 38.9 (8.5) | 42.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black, Non-Hispanic | 2 | 2 | 4
  Race/Ethnicity: White, Hispanic | 8 | 6 | 14
  Race/Ethnicity: White, Non-Hispanic | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS-5)
Description: The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders v5 (DSM-5) criteria for PTSD. Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms.Subscale scores are calculated by summing severity scores for items in the following PTSD symptom clusters: re-experiencing, avoidance, negative alterations in cognitions and mood, and hyperarousal. Scores ≥ 25 indicate a probable diagnosis of PTSD. Scores range from 0 to 80. Change in score will be reported.
Time Frame: Baseline and at about 45 days (1 month follow-up visit)
Population: Intent to treat analysis were completed in the total sample (n=21; CBD = 11, Placebo = 10).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cannabidiol (CBD) | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline | 42.8 (2.3) | 42.9 (2.2)
  1-Month Follow-Up | 15.2 (2.6) | 10.1 (2.6)

2. Primary Outcome: Posttraumatic Stress Disorder Checklist (PCL-5)
Description: The PCL-5 is a 20-item self-report measure update of the PCL designed to assess PTSD symptoms as defined by the DSM-5. The PCL-5 evaluates how much participants have been bothered by PTSD symptoms in the past week (for all assessments during treatment) or the past two weeks (all other assessment time points) as a result of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 "not at all") to 4 ("extremely). Scores range from 0 to 80 with a higher score indicating that subjects have been bothered more by PTSD symptoms. Change in score will be reported.
Time Frame: Baseline and at about 45 days (1 month follow-up visit)
Population: Intent to treat analysis were completed in the total sample (n=21; CBD = 11, Placebo = 10).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cannabidiol (CBD) | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline | 50.8 (0.9) | 52.1 (0.9)
  1-Month Follow-Up | 19.97 (7.6) | 27.3 (8.1)

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the diagnostic criteria for Diagnostic Statistical Manual of Mental Disorders - Major Depressive Disorder (DSM MDD). Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores on all items are summed to obtain a total severity score between 0 and 27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (>19). Change in score is reported.
Time Frame: Baseline and at about 45 Days (1 month follow-up visit)
Population: Intent to treat analysis were completed in the total sample (n=21; CBD = 11, Placebo = 10).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cannabidiol (CBD) | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline | 14.6 (0.5) | 15.5 (0.5)
  1-Month Follow-Up | 5.4 (2.4) | 7.3 (2.4)

ADVERSE EVENTS:
Time Frame: Enrolled participants were monitored for AEs at Interim Assessment 1 (PE Session 1), Interim Assessment 2 (PE Session 5), Interim Assessment 3 (PE Session 10), and at the 1-month follow-up.
Description: AEs were assessed/monitored using standardized procedures. At each assessment period, participants were asked "Have you experienced any changes for the worse since your last visit?" Reported events were documented by the research team member. Participants were asked about the temporal nature (start/stop date), severity, impact on functioning, and whether the event is study-related. AEs were reviewed during biweekly study meetings to ensure reliable coding and participant safety.
Arm/Group | Cannabidiol (CBD) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 10/11 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (CBD) (N=11) | Placebo (N=10)
Gastrointestinal Issues (Gastrointestinal disorders) | 4 (4) | 2 (2) — diarrhea, cramps, nausea
Emotional Problems (Psychiatric disorders) | 3 (3) | 1 (1) — increased emotional distress, anger, emotional numbness
Fatigue (Psychiatric disorders) | 2 (2) | 3 (3) — fatigue attributed to prolonged exposure
Sleep Disturbance (Psychiatric disorders) | 4 (4) | 0 (0) — increased nightmares and increased difficulty falling/staying asleep
Sensation from study drug (General disorders) | 0 (0) | 2 (2) — instant burning/warm sensation when taking study drug
Appetite Increase (General disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0) — drowsiness attributed to study drug
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Increased joint pain in knee attributed to stopping medication following participation
Physiological Arousal (Psychiatric disorders) | 1 (1) | 0 (0) — Increased physiological arousal attributed to prolonged exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT05132699/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT05132699/ICF_000.pdf